CLINICAL TRIAL: NCT03943836
Title: Reducing Anxiety in Pediatric Dental Patient Through Passive Musical Therapy
Brief Title: Reducing Anxiety in Pediatric Dental Patients Through Passive Music Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: PI, who was a Resident, graduated, and the project was not pursued further.
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Brett Thomas Chiquet, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HSC-DB-19-0220
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Anxiety, Dental
Keywords: Dental Anxiety; Pediatric dentistry
MeSH Terms: conditions — Anxiety Disorders | interventions — Music Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music Group (Experimental): Patients listen to music
  Interventions: Behavioral: Music
- No Music group (No Intervention): Patients do not listen to music

INTERVENTIONS:
Behavioral: Music — Patients in the music group will listen to classical music during their dental procedure.
  Arms: Music Group

SUMMARY:
The purpose of this study is to determine if passive music listening decreases anxiety in patients undergoing dental procedures and if the effects of music therapy are influenced by gender, age, and amount or type of dental treatment needed.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Physical Status Classification System I (ASA I) I and American Society of Anesthesiologists Physical Status Classification System II (ASA II)
* Patient needs restorative procedure (with or without local anesthesia or nitrous oxide)
* Received previous dental restorative treatment (detected via visual or radiographic evidence of previous restoration - no additional radiographs will be exposed for this study; exposed radiographs will be previously obtained, as needed,for comprehensive or periodic dental reasons)

Exclusion Criteria:

* Patients with hearing impairments
* Uncooperative patients at examination appointment (detected by Frankl behavior score of 1 or 2)

Ages: 9 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Anxiety as assessed by the Pediatric 7 question survey | baseline
  The total score ranges from 7-49, with lower scores indicating less anxiety.
Anxiety as assessed by the Pediatric 7 question survey | immediately after the dental procedure (within 5 minutes after procedure)
  The total score ranges from 7-49, with lower scores indicating less anxiety.
Parent's prediction of child's anxiety in the dental office as assessed by survey | baseline
  The total score ranges from 0-10. A lower score indicates less anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Ly, DDS, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No